CLINICAL TRIAL: NCT02926560
Title: Study Medication Adherence and Its Determinants in Chronic Disease Through the Example of Methotrexate in Chronic Inflammatory Rheumatism
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2015/CGV-02
Record Dates: First submitted 2016-09-16; First posted 2016-10-06 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Rheumatic Diseases
Keywords: Chronic inflammatory rheumatism
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The aim of this study is

1) To describe the level and determinants of methotrexate adherence in patients with chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis and psoriatic arthritis) in the department of rheumatology in the Nîmes University Hospital

ELIGIBILITY:
Inclusion Criteria:

* treated by methotrexate
* patients with chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis and psoriatic arthritis)

Exclusion Criteria:

* methotrexate for other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis and psoriatic arthritis) treated by methotrexate in the department of rheumatology in the Nîmes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Measure= Morisky scale | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Gaujoux-Viala, MD,PhD, Principal Investigator — CHU Nîmes
Locations (1):
- CHU Nîmes, Nîmes, Gard, France